

Certain information within this clinical study report has been redacted (ie, specific content is masked irreversibly from view with a black bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).



#### STATISTICAL ANALYSIS PLAN

STUDY NUMBER: TAK-385/CCT-002

A Multicenter, Randomized, Double-Blind, Parallel-Group, Phase 3 Study to Evaluate the Efficacy and Safety of Oral TAK-385 40 mg compared with Leuprorelin in the Treatment of Uterine Fibroids

#### PHASE 3

Version: Final

Date: 1 AUG 2017

# Prepared by:



Based on:

Protocol Version: Original

Protocol Date: 24 November 2015

#### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.

# 1.1 Approval Signatures

Electronic signatures can be found on the last page of this document.

#### 2.0 TABLE OF CONTENTS 10 1.1 2.0 List of In-Text Figures ......4 3.0 LIST OF ABBREVIATIONS......5 40 4.1 4.2 4.3 4.4 5.0 5.1 5.2 53 6.0 DETERMINATION OF SAMPLE SIZE ......12 7.0 7.1 General Principles 13 7.2 7.3 7.3.1 7.3.2 Screen Failures 19 7.3.3 7.3.4 7.3.5 Protocol Deviations 21 7.3.6 Analysis Sets 22 7 4 7.5

| TAK-385/0<br>Statistical | CCT-002<br>Analysis Plan | Page 4 of 48<br>1 AUG 2017 |
|---|---|---|
| 7.6 | Medication History and Concomitant Medications | 25 |
| 7.7 | Study Drug Exposure and Compliance | 25 |
| 7.8 | Efficacy Analysis | |
| 7. | 8.1 Primary Efficacy Endpoint(s) | 26 |
| 7. | 8.2 Secondary Efficacy Endpoint(s) | 28 |
| 7. | 8.3 Additional Efficacy Endpoint(s) | 30 |
| 7.9 | Pharmacokinetic/Pharmacodynamic Analysis | 32 |
| 7. | 9.1 Pharmacokinetic Analysis | 32 |
| 7. | 9.2 Pharmacodynamic Analysis | 32 |
| 7.10 | Other Outcomes | |
| 7.11 | Safety Analysis | 33 |
| 7. | 11.1 Adverse Events | 33 |
| 7. | 11.2 Clinical Laboratory Evaluations | 38 |
| 7. | 11.3 Vital Signs | 40 |
| 7. | 11.4 12-Lead ECGs | 41 |
| 7. | 11.5 Other Observations Related to Safety | 41 |
| 7.12 | Interim Analysis | 43 |
| 7.13 | Changes in the Statistical Analysis Plan | 43 |
| 8.0 R | EFERENCES | 48 |
| LIST OF | IN-TEXT FIGURES | |
| Figure 4 | Schematic of Study Design | 9 |

#### 3.0 LIST OF ABBREVIATIONS

AE adverse event

AESI adverse event of special interest

ALP alkaline phosphatase
ALT alanine aminotransferase
AST aspartate aminotransferase

AUC area under the blood concentration-time curve

BAP bone specific alkaline phosphatase

BMD bone mineral density
BMI body mass index
BUN blood urea nitrogen

C<sub>max</sub> maximum observed plasma concentration

CRF case report form

CRO contract research organization

CT computed tomography

DXA dual-energy x-ray absorptiometry

E<sub>2</sub> estradiol

ECG electrocardiogram

eCRF electronic case report form

FAS full analysis set

FDA Food and Drug Administration

Fe iron

FSH follicle-stimulating hormone
GCP Good Clinical Practice
GGT gamma glutamyl transferase
GLDH glutamate dehydrogenase
GnRH gonadotropin-releasing hormone
hCG human chorionic gonadotropin

HCT hematocrit

HDL high density lipoprotein

HGB hemoglobin

ICH International Conference on Harmonisation

INN international non-proprietary name
INR international normalized ratio
IRB institutional review board

IUDintrauterine deviceLDHlactate dehydrogenaseLDLlow density lipoproteinLFTliver function testLHluteinizing hormone

MedDRA Medical Dictionary for Regulatory Activities

MHRA Medicines and Healthcare products Regulatory Agency

MRI magnetic resonance imaging

NILM negative for intraepithelial lesion or malignancy

NRS numerical rating scale

NSAIDs non-steroidal anti-inflammatory drugs

NTELOP N-telopeptide P progesterone

PBAC pictorial blood loss assessment chart

P-gp P-glycoprotein
PGx pharmacogenomics

PMDA Pharmaceuticals and Medical Devices Agency

PPS per protocol set
PT preferred term
PTE Pretreatment event
QOL quality of life

Run-in AE run-in adverse event

RBC red blood cell

SAE serious adverse event
SAP statistical analysis plan
SC subcutaneous(ly)

SERM selective estrogen receptor modulator

SOC system organ class

SUSARs suspected unexpected serious adverse reactions

TBA total bile acid

TEAE treatment-emergent adverse event

TPC Takeda Pharmaceutical Company Limited UFS-QOL uterine fibroid symptom and quality of life

ULN upper limit of normal WBC white blood cell

WHO World Health Organization

WPAI:GH Work Productivity and Activity Impairment Questionnaire:General Health

#### 4.0 OBJECTIVES

#### 4.1 Primary Objectives

The primary objective of this study is to evaluate the efficacy of TAK-385 40 mg administered orally once daily for 12 weeks, compared with leuprorelin injection (once/4 weeks, 1.88 mg or 3.75 mg subcutaneously [SC]/time) in subjects with uterine fibroids.

# 4.2 Secondary Objectives

The secondary objective of this study is to evaluate the efficacy and safety of TAK-385 40 mg administered orally once daily for 24 weeks, compared with leuprorelin injection (once/4 weeks, 1.88 mg or 3.75 mg SC/time) in subjects with uterine fibroids.

## 4.3 Additional Objectives

An additional objective of this study is to evaluate the pharmacodynamic effect, which is blood concentrations of luteinizing hormone (LH), follicle-stimulating hormone (FSH), estradiol (E<sub>2</sub>), and progesterone (P).

#### 4.4 Study Design

An overview of the study design is shown in Figure 4

#### 4.4.1 Study Population and Design

This is a phase 3, multicenter, randomized, double-blind, parallel-group, non-inferiority study to evaluate the efficacy and safety of TAK-385 compared with leuprorelin injection (once/4 weeks, 1.88 mg or 3.75 mg SC/time) in premenopausal subjects ≥ 20 years of age with symptomatic uterine fibroids. The primary objective is to evaluate the efficacy of TAK-385 40 mg administered orally once daily for 12 weeks. The secondary objective is to evaluate the efficacy and safety of TAK-385 40 mg administered orally once daily for 24 weeks. In addition, the pharmacodynamics of continuous oral administration of TAK-385 40 mg for 24 weeks is to be assessed.

Subjects must be diagnosed to have uterine fibroids as confirmed by transvaginal ultrasound or other methods, and have symptoms of menorrhagia (the total pictorial blood loss assessment chart [PBAC] score of  $\geq$  120 for the entire menstrual cycle immediately before VISIT 3). The total number of subjects to be randomized under double-blind conditions is 288 (144 subjects each for the TAK-385 40 mg group or leuprorelin group).

After signing the informed consent form, subjects will start recording in the patient diary from the day of VISIT 1. During the period between VISIT 2 and VISIT 3, in which subjects must experience 1 menstrual cycle, the baseline values for the efficacy evaluation, including PBAC scores and pain symptoms (baseline PBAC score: the total PBAC score for the entire menstrual cycle immediately before VISIT 3) will be collected. Subjects should record in the patient diary every day until the end of study drug administration. VISIT 2 should be between the first and

fifth day of the first menstruation after VISIT 1. The study drug (TAK-385 placebo and leuprorelin placebo) will be administered under single-blind conditions from the day of VISIT 2 to the day before VISIT 3. VISIT 3 should be between the first and fifth day of the second menstruation after VISIT 1. From VISIT 3 to 10, subjects will receive study drug (TAK-385 and leuprorelin placebo, or TAK-385 placebo and leuprorelin) in a double blind manner. Subjects should try to visit the study site during the morning in a fasted state and before taking the TAK-385 tablet.

The study consists of Screening of approximately 1 to 6 weeks, a Run-in period of 3 to 6 weeks, a Treatment period of 24 weeks, and a Follow-up period of 4 weeks. The total period of study participation is approximately 32 to 40 weeks. If the recovery of the first post-treatment menstruation is not observed by the visit at the end of the Follow-up (VISIT 11), the subject will undergo further follow-up using possible means such as by telephone interview, until the recovery of the first post-treatment menstruation is observed. During the course of this study, subjects will visit the study site to undergo the designated examinations and evaluations at each visit, every 2 weeks for a month after the initiation of study drug administration (VISIT 3) under double-blind conditions, and monthly thereafter.

## 4.4.2 Dose Level and Regimen

At VISIT 3, subjects will be randomized in a 1:1 ratio to either the TAK-385 40 mg group or leuprorelin group. Study drug (TAK-385 40 mg + leuprorelin placebo or TAK-385 placebo + leuprorelin) will be administered in a double-dummy method from the day of VISIT 3 to the day before VISIT 10 (or until early termination) under double-blind conditions.

The investigator or subinvestigator will decide the dosage of leuprorelin at VISIT 2 in accordance with the approved dosage and administration, considering the body weight and symptoms of the individual subject. Leuprorelin (or leuprorelin placebo) should be administered SC (injection) once every 4 weeks using the same dose throughout the Run-in and Treatment.

TAK-385 (or TAK-385 placebo) will be administered daily as a single oral dose before breakfast.

Figure 4 Schematic of Study Design



#### 5.0 ANALYSIS ENDPOINTS

#### 5.1 Primary Endpoint

1) Efficacy:

Proportion of subjects with a total PBAC score of < 10 from Week 6 to 12

# 5.2 Secondary Endpoints

- 1) Efficacy:
- Proportion of subjects with a total PBAC score of < 10 (from Week 2 to 6, from Week 18 to 24, and for 6 weeks before the final dose of study drug)
- Myoma volumes (Week 2, 4, 8, 12 and 24)

Note: Only the largest myoma among those measurable at VISIT 1 will be measured throughout the study.

- Uterine volumes (Week 2, 4, 8, 12 and 24)
- Hemoglobin (HGB) (Week 4, 8, 12, 16, 20, 24 and Follow-up)
- Numerical Rating Scale (NRS) score (from Week 6 to 12, from Week 2 to 6, from Week 18 to 24, and for 6 weeks before the final dose)
- Uterine fibroid symptom and QOL (UFS-QOL) score (Week 4, 8, 12, 16, 20, 24 and Follow-up)
- 2) Safety:
- Adverse events (AEs), vital signs, weight, standard 12-lead electrocardiogram (ECG), clinical laboratory tests, bone mineral density (BMD), biochemical bone metabolism markers (serum N-telopeptide [NTELOP] and bone specific alkaline phosphatase [BAP])

#### 5.3 Additional Endpoints

- 1) Efficacy:
- Hematocrit (HCT), serum iron (Fe), and serum ferritin (Week 4, 8, 12, 16, 20, 24 and Follow-up)
- Use of analgesic medications during the Treatment (from Week 6 to 12, from Week 2 to 6, from Week 18 to 24, and for 6 weeks before the final dose)
- Work Productivity and Activity Impairment Questionnaire:General Health (WPAI:GH) (Week 2, 4, 8, 12 and 24)
- 2) Safety:
- Period from the last dose of study drug to return of menstrual cycles

3) Pharmacodynamic effects:

LH, FSH,  $E_2$  and P (Week 2, 4, 8, 12, 16, 20, 24 and Follow-up)

#### 6.0 DETERMINATION OF SAMPLE SIZE

## Justification of Sample size

In a clinical study of ulipristal acetate (already approved in Europe) compared with leuprorelin conducted overseas, the proportion of subjects with a total PBAC score of < 75 for 28 days before Week 13 was 89.1% in the TAP-144-SR (1M) 3.75 mg group, and the proportion of subjects with a total PBAC score of  $\le 2$  for 28 days before Week 13 was 80.4%.

In TAK-385 phase 2 study in the treatment of uterine fibroids, the point estimate (and corresponding 2-sided 95% confidence interval) of the proportion of subjects with a total PBAC score of < 10 from Week 6 to 12 was 83.6% (71.2%, 92.2%) in the TAK-385 40 mg group.

Based on the results of the above 2 studies, the proportions of subjects with a total PBAC score of < 10 from Week 6 to 12 in both TAK-385 40 mg group and leuprorelin group are estimated to be 83.6%.

Under this assumption, a sample size of at least 129 subjects per group will provide  $\geq 90\%$  power to demonstrate non-inferiority at 1-sided 0.025 level of significance, using a non-inferiority margin of 15% (nQuery Advisor 6.01).

Based on the above, a sample size of 129 subjects per group (258 subjects in total) is planned as the number of evaluable subjects. Assuming that approximately 10% of subjects will not be evaluable for the primary endpoint, 144 subjects are to be randomized to each group, for a total of 288 subjects.

#### Justification of non-inferiority margin

As the result of the TAK-385 phase 2 study in the treatment of uterine fibroids, the point estimate (and corresponding 2-sided 95% confidence interval) of the difference in the proportion of subjects with a total PBAC score of < 10 from Week 6 to 12 was 83.6% (73.9%, 93.4%) between the TAK-385 40 mg group and Placebo group. Assuming that leuprorelin has comparable effect to TAK-385 40 mg, the non-inferiority margin of 15% is considered smaller than the smallest effect size that leuprorelin would be reliably expected to have.

#### 7.0 METHODS OF ANALYSIS AND PRESENTATION

# 7.1 General Principles

All statistical analyses will be conducted using SAS® Version 9.2, or higher.

A statistical test for the primary endpoint will be reported as 1-sided and will be assessed at  $\alpha$ =0.025 significance level and all confidence intervals will be reported as 2-sided unless otherwise stated. P-values will be rounded to 4 decimal places prior to assessment of statistical significance.

Means and medians will be presented to 1 more decimal place than the recorded data. The standard deviations (SDs) will be presented to 2 more decimal places than the recorded data. Confidence intervals about a parameter estimate will be presented using the same number of decimal places as the parameter estimate.

Where appropriate, variables will be summarized descriptively by study visit. For the categorical variables, the count and proportions of each possible value will be tabulated by treatment group. The denominator for the proportion will be based on the number of subjects who provided non-missing responses to the categorical variable. For continuous variables, the number of subjects with non-missing values, mean, median, SD, minimum, and maximum values will be tabulated. Confidence intervals for continuous variables will be calculated based on t-statistics and ones for categorical variables will be based on Wald confidence intervals without using any model, unless otherwise stated.

### 7.1.1 Study Definitions

Duration of exposure to double-blind study drug (days):

Date of last dose of double-blind study drug - date of first dose of double-blind study drug + 1

Double-blind study drug compliance (%):

Number of TAK-385 blinded drugs taken/duration of exposure to TAK-385 blinded drug \* 100 (rounded to 1 decimal places )

Disease duration (years):

((year of informed consent\*12 + month of informed consent) –(year of first defined diagnosis of uterine fibroids\*12 + month of first defined diagnosis of uterine fibroids))/12 (rounded to 1 decimal places)

Maximum drug holidays (days):

Maximum number of consecutive days on which the subject does not take the TAK-385 blinded drug for the treatment period

Total PBAC score from Week 6 to 12

Total PBAC score from Day 43 to earlier of Day 84 or Follow-up Day 3. Similarly, Total PBAC score from Week 2 to 6 and from Week 18 to 24 will be defined as

those from Day 15 to earlier of Day 42 or Follow-up Day 3 and from Day 127 to earlier of Day 168 or Follow-up Day 3, respectively.

Total PBAC score for 6 weeks before the final dose of study drug Total PBAC score for the last 42 days of the treatment

NRS score from Week 6 to 12

Average NRS score from Day 43 to earlier of Day 84 or Follow-up Day 3.

Similarly, NRS score from Week 2 to 6 and from Week 18 to 24 will be defined as average NRS score from Day 15 to earlier of Day 42 or Follow-up Day 3 and from Day 127 to earlier of Day 168 or Follow-up Day 3, respectively.

NRS score for 6 weeks before the final dose

Average NRS score for the last 42 days of the treatment

Total PBAC at baseline

Total PBAC score from first day of menstrual period confirmed at Visit 2 to a day prior to menstrual period confirmed at Visit 3

NRS score at baseline

Average NRS score from first day of menstrual period confirmed at Visit 2 to a day prior to menstrual period confirmed at Visit 3

Use of analgesic medications during the treatment from Week 6 to 12

((number of days with analgesic medications use between Day 43 and earlier of Day 84 or Follow-up Day 3)/(number of days with available data between Day 43 and earlier of Day 84 or Follow-up Day 3))\*100 (rounded to 1 decimal places)

Similarly, use of analgesic medications during the treatment from Week 2 to 6 and from Week 18 to 24 will be defined as proportion of days with analgesic use between Day 15 and earlier of Day 42 or Follow-up Day 3 and between Day 127 and earlier of Day 168 or Follow-up Day 3, respectively.

Use of analgesic medications during the Treatment for 6 weeks before the final dose ((number of days with analgesic medications use for the last 42 days of the treatment)/(number of days with available data for the last 42 days of the treatment))\*100 (rounded to 1 decimal places)

Proportion of subjects with a total PBAC score of < 10 from Week 6 to 12:

((number of subjects with a total PBAC score of less than 10 from Week 6 to 12)/( number of subjects with available PBAC score from Week 6 to 12))\*100 (rounded to 1 decimal places)

Myoma volumes

 $D1*D2*D3*\pi/6 \text{ (cm}^3)$ 

Uterine volumes will be similarly calculated.

Definitions of D1, D2 and D3 are shown in protocol.

**Duration of Menstruation Recovery** 

Date of menstruation recovery - date of last dose of double-blind study drug Oral iron preparation

The drug with the following drug code of WHODD: 00023503001, 00023505001, 00023520001, 00023550009, 00023550074, 90059601001

### 7.1.2 Definition of Study Days

When calculating Study Day relative to a reference date (ie, date of first dose of double-blind study drug [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

When calculating Follow-up Day relative to a reference date (ie, date of last dose of double-blind study drug [Follow-up Day 0]), it will be calculated as: date of observation - reference date. Hence, reference day is always Follow-up Day 0.

# 7.1.3 Definition of Study Visit Windows

All evaluable data (ie, non-missing and acceptable according to the Handling Rules for Analysis Data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used.

#### Transvaginal ultrasound and WPAI

| X7: :4 | Scheduled Study Day | Time Inter | val (days) |
|----------|---------------------|------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -80 - 1 | |
| Week 2 | Study Day: 15 | 2 - 22 | < 4 |
| Week 4 | Study Day: 29 | 23 - 43 | < 4 |
| Week 8 | Study Day: 57 | 44 - 71 | < 4 |
| Week 12 | Study Day: 85 | 72 - 127 | < 4 |
| Week 24 | Study Day: 169 | 128 – 183 | < 4 |

Anemia-related measurements (Hemoglobin [HGB], Hematocrit [HCT], Serum Fe, and Serum Ferritin) and UFS-QOL score

| Visit | Scheduled Study Day | Time Interval (days) |
|-------|---------------------|----------------------|
|-------|---------------------|----------------------|

| | (days) | Study Day | Follow-up Day |
|-----------|-------------------|-----------|---------------|
| Baseline | Study Day: 1 | -80 - 1 | |
| Week 4 | Study Day: 29 | 2 – 43 | < 4 |
| Week 8 | Study Day: 57 | 44 – 71 | < 4 |
| Week 12 | Study Day: 85 | 72 – 99 | < 4 |
| Week 16 | Study Day: 113 | 100 – 127 | < 4 |
| Week 20 | Study Day: 141 | 128 – 155 | < 4 |
| Week 24 | Study Day: 169 | 156 – 183 | < 4 |
| Follow-up | Follow-up Day: 28 | 2 <= | 4 – 42 |

# Clinical laboratory tests (except bile acid (total bile acid [TBA]) and glutamate dehydrogenase (GLDH)) and vital sign and weight

| ****** | Scheduled Study Day | Time Interval (days) | |
|-----------|---------------------|----------------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -80 - 1 | |
| Week 4 | Study Day: 29 | 2 – 43 | < 15 |
| Week 8 | Study Day: 57 | 44 – 71 | < 15 |
| Week 12 | Study Day: 85 | 72 – 99 | < 15 |
| Week 16 | Study Day: 113 | 100 - 127 | < 15 |
| Week 20 | Study Day: 141 | 128 – 155 | < 15 |
| Week 24 | Study Day: 169 | 156 – 183 | < 15 |
| Follow-up | Follow-up Day: 28 | 2 <= | 15 – 42 |

# Pharmacodynamic measurements

| <b>X</b> 7: :4 | Scheduled Study Day | Time Inter | val (days) |
|----------------|---------------------|------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -80 - 1 | |
| Week 2 | Study Day: 15 | 2 - 22 | < 4 |
| Week 4 | Study Day: 29 | 23 - 43 | < 4 |
| Week 8 | Study Day: 57 | 44 – 71 | < 4 |
| Week 12 | Study Day: 85 | 72 – 99 | < 4 |
| Week 16 | Study Day: 113 | 100 – 127 | < 4 |

| 77° ' | Scheduled Study Day | Time Interval (days) | |
|-----------|---------------------|----------------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Week 20 | Study Day: 141 | 128 – 155 | < 4 |
| Week 24 | Study Day: 169 | 156 – 183 | < 4 |
| Follow-up | Follow-up Day: 28 | 2 <= | 4 – 42 |

# Clinical laboratory tests (TBA and GLDH)

| ¥7° °, | Scheduled Study Day | Time Interval (days) | |
|-----------|---------------------|----------------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -80 - 1 | |
| Week 2 | Study Day: 15 | 2 – 22 | < 15 |
| Week 4 | Study Day: 29 | 23 - 43 | < 15 |
| Week 8 | Study Day: 57 | 44 – 71 | < 15 |
| Week 12 | Study Day: 85 | 72 – 99 | < 15 |
| Week 16 | Study Day: 113 | 100 – 127 | < 15 |
| Week 20 | Study Day: 141 | 128 – 155 | < 15 |
| Week 24 | Study Day: 169 | 156 – 183 | < 15 |
| Follow-up | Follow-up Day: 28 | 2 <= | 15 – 42 |

# 12-lead ECG

| <b>X</b> 74 | Scheduled Study Day | Time Interval (days) | |
|-------------|---------------------|----------------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -80 - 1 | |
| Week 24 | Study Day: 169 | 2 - 183 | < 15 |
| Follow-up | Follow-up Day: 28 | 2 <= | 15 – 42 |

# Biochemical bone metabolism markers and BMD

| ******* | Scheduled Study Day | Time Inter | val (days) |
|----------|---------------------|------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -80 - 1 | |

| *** */ | Scheduled Study Day | Time Inter | val (days) |
|---------|---------------------|------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Week 12 | Study Day: 85 | 2 – 127 | < 15 |
| Week 24 | Study Day: 169 | 128 - 183 | < 15 |

# 7.1.4 Methods for Handling Missing Data

All available efficacy and safety data will be included in data listing and tabulations. No imputation of values for missing data will be performed unless otherwise specified.

- For UFS-QoL and WPAI, published scoring manuals and guidelines will be used to calculate UFS-QoL and WPAI scale scores and handle missing data (see Appendix 3 and 4, respectively).
- For myoma or uterus volume, if D1 and D2 of the myoma or uterus are present but D3 is missing, then the volume will be calculated as D1\*D2\*D2\* $\pi$ /6 (cm<sup>3</sup>).
- For LH, FSH, E<sub>2</sub>, P and clinical laboratory tests, values less than the lower limit of quantification will be treated as zero when calculating the descriptive statistics.
- Disease duration with first diagnosis date of uterine fibroid that are completely or partially missing will be derived as follows:
  - 1. If the year is missing, then the disease duration will be treated as missing.
  - 2. If the year is present but the month is missing, then the month will be treated as January for the calculation.

# 7.2 Analysis Sets

Refer to the Handling Rules for Analysis Data.

## 7.3 Disposition of Subjects

# 7.3.1 Study Information

Analysis Set: All Subjects Who Signed the Informed Consent Form

**Analysis** 

Variable(s): Date first subject signed informed consent form

Date of last subject's last visit/contact

MedDRA version

WHO Drug version

SAS version used for creating the datasets

Analytical

Method(s): (1) Study Information

Study information shown in the analysis variables section will be

provided.

#### 7.3.2 Screen Failures

Analysis Set: All Subjects Who Were Not Randomized

Analysis

Variable(s): Age (years) [20<= - <30, 30<= - <40, 40<= -

<50, 50<= -<=Max

Analytical

Method(s): (1) Screen Failures

Frequency distributions for categorical variables and descriptive

statistics for continuous variables will be provided.

# 7.3.3 Subject Eligibility

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): Eligibility status [Eligible for Randomization, Not

Eligible for Randomization]

Primary Reason for Subject Not [Death, Adverse Event, Screen

Being Eligible Failure, Protocol Deviation, Lost to

Follow-up, Withdrawal by Subject,

Study Terminated by Sponsor,

Pregnancy, Other]

Analytical

Method(s): (1) Eligibility for Randomization

Frequency distributions will be provided. When calculating

percentages for the primary reasons for subject not being eligible,

the total number of ineligible subjects will be used as the

denominator.

# 7.3.4 Number of Subjects Randomized by Site and Treatment Group

Analysis Set: Randomized Set

Analysis

Variable(s): Randomization status [Randomized]

Stratum: Site [Site numbers will be used as

categories]

Analytical

Method(s): (1) Number of Subjects Randomized by Site and Treatment Group

Frequency distribution will be provided for each stratum by treatment

group and overall.

# 7.3.5 Disposition of Subjects

Analysis Set: Randomized Set

Analysis Double-blind study drug

Variable(s): administration status [Randomized but Not Treated]

Reason for not being treated [Death, Adverse Event, Protocol

Deviation, Lost to Follow-up, Withdrawal by Subject, Study

Terminated by Sponsor,

Pregnancy, Lack of Efficacy, Bone Mineral Density Loss, Recovery Leading to Surgery, Reduction of

HGB Concentration, Other]

Double-Blind Study Drug [Completed Study Drug,

Completion Status Prematurely Discontinued Study

Drug]

Reason for Discontinuation of

Study Drug

[Death, Adverse Event, Protocol

Deviation, Lost to Follow-up, Withdrawal by Subject, Study

Terminated by Sponsor,

Pregnancy, Lack of Efficacy, Bone Mineral Density Loss, Recovery Leading to Surgery, Reduction of

HGB Concentration, Other]

Completion Status of the Follow- [Completed Follow-up Period,

up Period Prematurely Discontinued Follow-

up Period]

Reason for Discontinuation of

the Follow-up Period

[Death, Adverse Event, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study

Terminated by Sponsor,

Pregnancy, Lack of Efficacy, Bone Mineral Density Loss, Recovery Leading to Surgery, Reduction of

HGB Concentration, Other]

### Analytical

Method(s): (1)

(1) Disposition of Subjects

Frequency distributions will be provided for each treatment group and overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

#### 7.3.6 Protocol Deviations

Analysis Set: Randomized Set

Analysis

Variable(s): Protocol Deviation [Major GCP Violations, Deviations of Protocol

Entry Criteria, Deviations of Discontinuation Criteria, Deviations Related to Treatment Procedure or Dose, Deviations Concerning Excluded Medication or Therapy, Deviations to

Avoid Emergency Risk]

Analytical

Method(s): (1) Protocol Deviations

Frequency distribution will be provided by treatment group and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several

deviations that can be classified into the same category will be counted only once.

### 7.3.7 Analysis Sets

Analysis Set: Randomized Set

Analysis

Variable(s): Handling of Subjects and Subject [Categories are based on the

Data specifications in Handling Rules

for Analysis Data]

**Analysis Sets** 

Full Analysis Set [Included]
Per Protocol Set [Included]
Safety Analysis Set [Included]

Analytical

Method(s): (1) Subjects Excluded from Analysis Sets

(2) Subject Data Excluded from Analysis Sets

(3) Analysis Sets

Frequency distributions will be provided by treatment group for (1) and (2), and by treatment group and overall for (3). For (1) and (2), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

# 7.4 Demographic and Other Baseline Characteristics

Analysis Set: Randomized Set

Analysis

Variable(s): Age (years)  $[20 \le -30, 30 \le -40,$ 

 $40 \le - <50, 50 \le - <= Max$ 

Height (cm)  $[Min \le -.. \le 150, 150 \le -.. \le 160,$ 

 $160 \le -170, 170 \le -180$ 

Weight (kg) at Baseline  $[Min \le -.. \le 50, 50 \le -.. \le 60,$ 

 $60 \le -80$ ,  $70 \le -80$ ,

| | $80 \le - \le Max$ |
|---|---|
| BMI (kg/m <sup>2</sup> ) at Baseline | [Min<= - <18.5, 18.5<= - <25.0, |
| | 25.0<= - <=Max] |
| Smoking Classification | [The subject has never smoked, |
| | The subject is a current smoker, |
| D' 4 E | The subject is an ex-smoker] |
| Birth Experience | [Yes, No] |
| Disease Duration (years) | [Min<= - <=1, 1< - <=3, 3< - <=5, |
| | 5 < - <= 10, 10 < - <= Max |
| Type of Uterine Fibroid | [X/ XI.] |
| Subserosal Fibroid<br>Intramural Fibroid | [Yes, No]<br>[Yes, No] |
| Submucosal Fibroid | [Yes, No] |
| Cervical Fibroid | [Yes, No] |
| Stopped Any Medications for | L / J |
| Uterine Fibroids | [Yes, No] |
| Type of Medication for Uterine | |
| Fibroid | [\$7] |
| GnRH Agonist<br>Herbal Medicine | [Yes]<br>[Yes] |
| Other Medicines for Uterine | [105] |
| Fibroids | [Yes] |
| Any Surgery for Uterine Fibroids | [Yes, No] |
| Volume of Myoma at Baseline | [Min<= - <=28, 28< - <=170, |
| (cm <sup>3</sup> ) | 170< - <=700, 700< - <=Max] |
| Volume of Uterus at Baseline | [Min<= - <=28, 28< - <=170, |
| $(cm^3)$ | 170< - <=700, 700< - <=Max] |
| PBAC Score at Baseline | [120<= - <200, 200<= - <500, |
| | 500<= - <=Max] |
| NRS Score at Baseline | [Min<= - <4, 4<= - <7, 7<= - |
| | <=Max] |
| UFS-QOL Score at Baseline | |
| Symptom Severity | [Min<= - <=25, 25< - <=50, |
| Concern | 50< - <=75, 75< - <=Max]<br>[Min<= - <=25, 25< - <=50, |
| Concern | 50< - <=75, 75< - <=Max] |
| Activities | [Min <= - <= 25, 25 < - <= 50, |
| | 50< - <=75, 75< - <=Max] |
| COMPINE | TODA A T |

| Energy/Mood | [Min<= - <=25, 25< - <=50, |
|---|---|
| | 50< - <=75, 75< - <=Max] |
| Control | [Min<= - <=25, 25< - <=50,<br>50< - <=75, 75< - <=Max] |
| Self-consciousness | [Min <= - <= 25, 25 < - <= 50, |
| | 50< - <=75, 75< - <=Max] |
| Sexual Function | [Min<= - <=25, 25< - <=50, |
| HRQL Total | 50< - <=75, 75< - <=Max]<br>[Min<= - <=25, 25< - <=50, |
| TINQL Total | 50 < - <= 75, 75 < - <= Max |
| HGB at Baseline (g/dL) | [Min<= - <10, 10<= - <12, 12<= - |
| | <=Max] |

HCT at Baseline (%)

Serum Fe at Baseline (µg/dL)

Serum Ferritin at Baseline (ng/mL)

Dosage of leuprorelin vial [1.88 mg, 3.75 mg]

Analytical

Method(s): (1

(1) Summary of Demographics and Baseline Characteristics
Frequency distributions for categorical variables and descriptive
statistics for continuous variables will be provided by treatment group
and overall.

# 7.5 Medical History and Concurrent Medical Conditions

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medical History

**Concurrent Medical Conditions** 

Analytical

Method(s): (1) Medical History by System Organ Class and Preferred Term

(2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided for each treatment group. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

# 7.6 Medication History and Concomitant Medications

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medication History

**Concomitant Medications** 

Analytical

Method(s): (1) Medication History by Preferred Medication Name

(2) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name

Frequency distributions will be provided for each treatment group. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that preferred medication name.

# 7.7 Study Drug Exposure and Compliance

Analysis Set: Safety Analysis Set

Analysis Duration of Exposure to Double-  $[1 \le - \le 14, 15 \le - \le 42,$ 

Variable(s): Blind Study Drug (days) 43<= - <=84, 85<= - <=168

 $169 \le - \le Max$ 

Double-Blind Study Drug [Min<= - <80, 80<= - <90, 90<= -

Compliance (%) <=Max]

Maximum Drug Holidays (days)  $[0, 1 \le -4, 4 \le -4]$ 

Exposure to Double-Blind [0, 1, 2, 3, 4, 5, 6]

leuprorelin vial (times)

Analytical

Method(s): (1) Study Drug Exposure and Compliance

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided by treatment group and overall.

7.8 Efficacy Analysis

# 7.8.1 Primary Efficacy Endpoint(s)

## 7.8.1.1 Primary Analysis

Analysis Set: Full Analysis Set

Analysis

Variable(s): Proportion of subjects with a total PBAC score of < 10 from Week 6 to

12

Analytical The point estimate and 2-sided 95% confidence interval of the proportion

Method(s): of subjects with a total PBAC score of < 10 from Week 6 to 12 will be

summarized by treatment group. The point estimate and 2-sided 95% confidence interval of the difference in the percentage will be calculated between TAK-385 40 mg group and leuprorelin group (TAK-385 40 mg group – leuprorelin group), using Farrington and Manning (FM) method. In addition, non-inferiority test using FM method with a non-inferiority margin of 15% will be conducted for the comparison between TAK-385 40 mg group and leuprorelin group. If the lower bound of the 95%CI is

greater or equal to the non-inferiority margin of -15%, then non-inferiority of TAK-385 40mg to leuprorelin will be concluded.

#### 7.8.1.2 Secondary Analysis

Analysis Set: Per Protocol Set

Analysis

Variable(s): Proportion of subjects with a total PBAC score of < 10 from Week 6 to

12

Analytical

Method(s): An analysis similar to the above "Primary analysis" will be performed

using the PPS to assess the robustness of the results.

### 7.8.1.3 Adjustments for Covariates

Analysis Set: Full Analysis Set

Analysis

Variable(s): Proportion of subjects with a total PBAC score of < 10 from Week 6 to

12

Covariate(s): PBAC Score at Baseline [120<= - <200, 200<= - <500,

 $500 \le - \le Max$ 

Analytical

Method(s): The difference between groups in the proportion of subjects with a total

PBAC score of < 10 from Week 6 to 12 will be analyzed using binomial regression with the identity link that includes treatment group and PBAC

score at baseline as independent categorical variable.

## 7.8.1.4 Examination of Subgroups

Analysis Set: Full Analysis Set

Analysis

Variable(s): Proportion of subjects with a total PBAC score of < 10 from Week 6 to

12

Subgroup(s): Age (years)  $[20 \le -30, 30 \le -40,$ 

 $40 \le - <50, 50 \le - <= Max$ 

BMI (kg/m<sup>2</sup>) at Baseline  $[Min \le -... \le 18.5, 18.5 \le -... \le 25.0,$ 

 $25.0 \le - \le Max$ 

PBAC Score at Baseline [120<= - <200, 200<= - <500,

 $500 \le - \le Max$ 

Birth Experience [Yes, No]

Volume of Uterus at Baseline [Min<= - <=28, 28< - <=170,

 $(cm^3)$  170< - <=700, 700< - <=Max]

Type of Uterine Fibroid

Subserosal Fibroid [Yes, No]
Intramural Fibroid [Yes, No]
Submucosal Fibroid [Yes, No]

Analytical

Method(s): (1) Descriptive Statistics

The point estimate and 2-sided 95% confidence interval of the proportion of subjects with a total PBAC score of < 10 from Week 6 to 12 will be summarized for above each subgroup by treatment group.

## 7.8.2 Secondary Efficacy Endpoint(s)

#### 7.8.2.1 *PBAC Score*

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): Proportion of subjects with a total PBAC score of < 10 from Week 2 to 6

Proportion of subjects with a total PBAC score of < 10 from Week 18 to

24

Proportion of subjects with a total PBAC score of < 10 for 6 weeks

before the final dose of study drug

Analytical

Method(s): For each variable, frequency will be summarized by treatment group.

The point estimate and 2-sided 95% confidence interval of the difference in the percentage will be calculated between TAK-385 40 mg group and leuprorelin group, using FM method with the non-inferiority margin of -15%. The confidence interval will be presented in a descriptive manner

and not for the purpose of statistical inference.

# 7.8.2.2 Myoma Volumes and Uterine Volumes

Analysis Set: Full Analysis Set

Analysis

Variable(s): Myoma volumes

Uterine volumes

Visit: Baseline, Week 2, 4, 8, 12 and 24

Analytical

Method(s): For each variable, descriptive statistics will be provided for the observed

values and the percent changes from baseline by treatment group for

each visit.

The mean differences in the percent changes from baseline between TAK-385 40 mg and leuprorelin group and the two-sided 95% confidence intervals will be provided.

# 7.8.2.3 Hemoglobin

Analysis Set: Full Analysis Set

Analysis

Variable(s): HGB (g/dL) [Min<= - <12, 12<= - <=Max]

Change from baseline on HGB  $[Min \le - <1, 1 \le - \le Max]$ 

(g/dL)

Subgroup(s): Oral iron preparation use at [Yes, No]

baseline

HGB at Baseline (g/dL)  $[Min \le - \le 12, 12 \le - \le Max]$ 

Visit: Baseline, Week 4, 8, 12, 16, 20, 24 and Follow-up

Analytical

Method(s): Summary statistics will be provided for the observed values and the

changes from baseline by treatment group for each visit.

The mean differences in the change from baseline between TAK-385 40 mg and leuprorelin groups and the two-sided 95% confidence

intervals will be provided for each visit.

For categorical variables, frequency will be summarized by treatment group for each visit. The differences in the percentage between TAK-385 40 mg and leuprorelin groups and the two-sided 95% confidence

intervals will be provided for each visit.

Additionally, the above mentioned analysis will also be conducted for

each subgroup.

#### 7.8.2.4 NRS Score

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): NRS score from Week 6 to 12

NRS score from Week 2 to 6 NRS score from Week 18 to 24

NRS score for 6 weeks before the final dose

Analytical

Method(s): For each variable, summary statistics will be provided by treatment

group. Two-sided 95% confidence interval of the difference will be

calculated between TAK-385 40 mg and leuprorelin group.

7.8.2.5 UFS-QOL Score

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): Symptom Severity

Concern Activities

Energy/Mood

Control

Self-consciousness Sexual Function HRQL Total

Visit: Baseline, Week 4, 8, 12, 16, 20, 24 and Follow-up

Analytical

Method(s): For each variable, descriptive statistics will be provided for the observed

values and the changes from baseline by treatment group for each visit. The mean differences in the observed values between TAK-385 40 mg and leuprorelin group and the two-sided 95% confidence intervals will

be provided for each visit.

#### 7.8.3 Additional Efficacy Endpoint(s)

7.8.3.1 Hematocrit, Serum Fe, and Serum Ferritin

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): HCT

Serum Fe

Serum ferritin

Visit: Baseline, Week 4, 8, 12, 16, 20, 24 and Follow-up

Analytical

Method(s): For each variable, summary statistics will be provided for the observed

values and the changes from baseline by treatment group for each visit.

# 7.8.3.2 Use of Analgesic Medications During the Treatment

Analysis Set: Full Analysis Set

Analysis

Variable(s): Use of analysesic medications during the Treatment from Week 6 to 12

Use of analyseic medications during the Treatment from Week 2 to 6 Use of analyseic medications during the Treatment from Week 18 to 24 Use of analyseic medications during the Treatment for 6 weeks before

the final dose

Analytical

Method(s): For each variable, summary statistics will be provided by treatment

group.

#### 7.8.3.3 WPAI:GH During the Treatment

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): Absenteeism

Presenteeism

Work productivity loss Activity impairment

Visit: Baseline, Week 2, 4, 8, 12 and 24

Analytical

Method(s): For each variable, summary statistics will be provided for the observed

values and the changes from baseline by treatment group for each visit. The mean differences in the observed values between TAK-385 40 mg and leuprorelin group and the two-sided 95% confidence intervals will

be provided for each visit.

# 7.8.3.4 *Amenorrhea (The subject with a total PBAC score of 0)*

Analysis Set: Full Analysis Set

Analysis

Variable(s): Proportion of subjects with a total PBAC score of 0 from Week 6 to 12

Proportion of subjects with a total PBAC score of 0 from Week 2 to 6 Proportion of subjects with a total PBAC score of 0 from Week 18 to 24 Proportion of subjects with a total PBAC score of 0 for 6 weeks before

the final dose of study drug

Analytical

Method(s): For each variable, frequency will be summarized by treatment group.

The point estimate and 2-sided 95% confidence interval of the difference in the percentage will be calculated between TAK-385 40 mg group and leuprorelin group, using FM method with the non-inferiority margin of -15%. The confidence interval will be presented in a descriptive manner

and not for the purpose of statistical inference.

# 7.9 Pharmacokinetic/Pharmacodynamic Analysis

#### 7.9.1 Pharmacokinetic Analysis

Not applicable

#### 7.9.2 Pharmacodynamic Analysis

7.9.2.1 LH, FSH,  $E_2$ , and P

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): LH

**FSH** 

 $E_2$ 

P

Visit: Baseline, Week 2, 4, 8, 12, 16, 20, 24 and Follow-up

Analytical

Method(s): For each variable, summaries (1) and (2) will be provided by treatment

group.

- (1) Summary of each variable and Change from Baseline by Visit Descriptive statistics for observed values for each visit and changes from baseline will be provided.
- (2) Case Plots
  Plots over time for each subject will be presented.

#### 7.10 Other Outcomes

Not applicable

## 7.11 Safety Analysis

#### 7.11.1 Adverse Events

# 7.11.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Treatment-emergent adverse event (TEAE)

Categories: Relationship to Study Drug [Related, Not Related]

Intensity [Mild, Moderate, Severe]

Analytical

Method(s): The following summaries will be provided for each treatment group.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 4) Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 6) Relationship of serious Treatment-Emergent Adverse Events to

- study drug (number of events, number and percentage of subjects)
- 7) Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

# Number of subjects

- Summaries for 2) and 6)
  - A subject with occurrences of TEAE in both categories (ie, Related and Not Related) will be counted once in the Related category.
- Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

Summaries other than 2), 3), and 6)
 A subject with multiple occurrences of TEAE will be counted only once.

#### Number of events

For each summary, the total number of events will be calculated.

# 7.11.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Categories: Intensity [Mild, Moderate, Severe]

Time of Onset (day) [1<= - <=28, 29<= - <=56, 57<= - <=84, 85<= - <=112, 113<= -

<=140, 141<= - <=168, 169<= -

 $\leq = Max$ 

Analytical

Method(s): The following summaries will be provided using frequency distribution

for each treatment group.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (10)Most Frequent Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (11)Most Frequent Non-Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Number of subjects

Summary tables other than (5), (6) and (9)
 A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT.
Percentages will be based on the number of subjects in the safety analysis set.

• Summary tables for (5) and (6)

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.

• Summary table for (9)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT.

When calculating percentages for each time interval, the number of subjects at risk (ie, subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

• Summary table for (10)

Most frequent TEAEs refer to PTs whose percentages are at least 5.0% in any one of the treatment groups.

• Summary table for (11)

Most frequent Non-Serious TEAEs refer to PTs whose percentages are at least 5.0% in any one of the treatment groups. If no Non-Serious TEAEs exceed a frequency of 5.0%, the frequency cutoff of 2.0% will be used instead. Percentages will be based on the number of subjects in the safety analysis set.

#### 7.11.1.3 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): Pretreatment event (PTE)

Analytical The following summaries will be provided using frequency distribution.

Method(s): PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term
- (2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

# 7.11.1.4 Displays of Run-in Adverse Events

Analysis Set: All Subjects Who Received Run-in Study Drug

Analysis

Variable(s): Run-in AE

Analytical The following summaries will be provided using frequency distribution.

Method(s): Run-in AEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Run-in Adverse Events by System Organ Class and Preferred Term
- (2) Drug-Related Run-in Adverse Events by System Organ Class and Preferred Term
- (3) Serious Run-in Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Number of subjects

A subject with multiple occurrences of run-in AE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of run-in AE within a PT will be counted only once in that PT.

### 7.11.2 Clinical Laboratory Evaluations

7.11.2.1 Hematology and Serum Chemistry

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Hematology

RBC Platelets WBC

WBC Differentials (Neutrophils, Eosinophils, Basophils, Lymphocytes,

Monocytes)

Serum Chemistry

ALT AST Lactate dehydrogenase

(LDH)

Gamma glutamyl Albumin Alkaline phosphatase

transferase (GGT) (ALP)

Bilirubin (Total Protein (Total Cholesterol (Total

bilirubin) protein) cholesterol)
High density Low density Triglycerides

lipoprotein (HDL) lipoprotein (LDL)

cholesterol cholesterol

Glucose HGB A1C Creatinine

Blood urea nitrogen Creatine kinase Urate

(BUN)

Sodium Potassium Chloride
Calcium Phosphate Magnesium

Bile acid (total bile Glutamate acid [TBA]) dehydrogenase

(GLDH)

Visit: Baseline, Week 2\*, 4, 8, 12, 16, 20, 24 and Follow-up

\*: only TBA and GLDH

Analytical

Method(s): For each variable, summaries (1) to (3) will be provided by treatment

group.

For applicable variables, summaries (4) and (5) will be provided by

treatment group.

(1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

- (2) Case Plots
  - Plots over time for each subject will be presented.
- (3) Summary of Shifts of Laboratory Test Results
  Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

  For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.
- (4) Number and Percentage of Subjects with Markedly Abnormal Values of Laboratory Parameters Overall frequency distributions of MAV during treatment period will be provided. If a laboratory parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.
- (5) Number and Percentage of Subjects with Elevated Liver Enzyme Laboratory Parameters Overall frequency distributions of elevated hepatic parameters during treatment period will be provided. Further details are given in Appendix.

#### 7.11.2.2 Urinalysis

Analysis Set: Safety Analysis Set

**Analysis** 

Variable(s): Protein [-, +-, 1+, 2+, 3+, 4+]

Glucose [-, 1+, 2+, 3+, 4+, 5+]

Occult blood [-, +-, 1+, 2+, 3+]
Bilirubin [-, +-, 1+, 2+, 3+]
Urabilina con [-, 1+, 2+, 3+]

Urobilinogen [+-, 1+, 2+, 3+]

Visit: Baseline, Week 4, 8, 12, 16, 20, 24 and Follow-up

Analytical

Method(s): For each variable, summaries (1) and (2) will be provided by treatment

group.

(1) Number of Subjects in Categories of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

(2) Summary of Shifts of Urine Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided. For each urine laboratory test, the laboratory values will be classified as "Normal" or " Abnormal " relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

# 7.11.3 Vital Signs

7.11.3.1 Vital Signs and Weight

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Systolic Blood Pressure

Diastolic Blood Pressure

Pulse Rate

Body temperature

Weight

Visit: Baseline, Week 4, 8, 12, 16, 20, 24 and Follow-up

Analytical

Method(s): For each variable, summaries (1) and (2) will be provided by treatment

group.

For applicable variables, summary (3) will be provided by treatment

group.

(1) Summary of Vital Signs Parameters and Weight and Change from

Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

- (2) Case Plots
  - Plots over time for each subject will be presented.
- (3) Number and Percentage of Subjects with Markedly Abnormal Values of Vital Signs Parameters Overall frequency distributions of MAV during treatment period will be provided. If a vital sign parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### 7.11.4 12-Lead ECGs

7.11.4.1 12-lead ECG

Analysis Set: Safety Analysis Set

Analysis

Variable(s): 12-lead ECG Interpretation [Within Normal Limits, Abnormal but not

Clinically Significant, Abnormal and

Clinically Significant]

Visit: Baseline, Week24 and Follow-up

Analytical

Method(s): For 12-lead ECG interpretation, summary (1) will be provided by

treatment group.

(1) Summary of Shift of 12-lead ECG Interpretation Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

#### 7.11.5 Other Observations Related to Safety

7.11.5.1 Bone Mineral Density and Biochemical Bone Metabolism Markers

Analysis Set: Safety Analysis Set

Analysis

Variable(s): T score  $[Min \le -\le -2.500]$ 

Bone Mineral Density (g/cm<sup>2</sup>)

Percent Change from baseline on Bone

 $[Min \le - <-7, -7 \le - <= Max]$ 

Mineral Density (%)

NTELOP (nmol BCE/L)

Bone Type Alkaline Phosphatase (µg/L)

Visit: Baseline, Week 12, 24

Analytical

Method(s): For each variable except T score, summaries (1), (3), and (4) will be provided by treatment group.

For T score, summary (2), (3), (4), and (5) will be provided by treatment group.

- (1) Summary of Parameters and percent Change from Baseline by Visit Descriptive statistics for observed values for each visit and percent changes from baseline will be provided.
  - For categorical variables, frequency will be summarized by treatment group for each visit.
- (2) Summary of Parameters and Change from Baseline by Visit Descriptive statistics for observed values for each visit and changes from baseline will be provided.
- (3) Case Plots

Plots over time for each subject will be presented.

- (4) Mean Plot with Standard Deviations
  - For T score, mean of observed values and changes from baseline will be plotted by visit.
  - For other variables, mean of observed values and percent changes from baseline will be plotted by visit.
- (5) Summary of Shift of T score
  Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

# 7.11.5.2 Return of Menstrual Cycles

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Duration of Menstruation Recovery (Days)

Analytical

Method(s): Summary (1) will be provided by treatment group.

(1) Summary of Duration of Menstruation Recovery

Descriptive statistics for observed values will be provided.

# 7.12 Interim Analysis

Not applicable

# 7.13 Changes in the Statistical Analysis Plan

Change from previous version are described in following table.

| Page | Previous version | Current version | Reason |
|---|---|---|---|
| 14 | 7.1.1 Study Definitions | 7.1.1 Study Definitions Oral iron preparation The drug with the following drug code of WHODD: 00023503001, 00023505001, 00023520001, 00023550009, 00023550074, 90059601001 | Specify the definition of Oral iron preparation based on blind review |
| 17 | 7.1.4 Methods for Handling Missing Data | 7.1.4 Methods for Handling Missing Data • For LH, FSH, E2, P and clinical laboratory tests, values less than the lower limit of quantification will be treated as zero when calculating the descriptive statistics. | Specify how to deal with value with lower limit of quantification for LH, FSH, E2, P and clinical laboratory |

| 23 | 7.4Demographic and Other<br>Baseline Characteristics<br>Other Medicines for<br>UterineFibroids | 7.4Demographic and Other<br>Baseline Characteristics<br>Other Medicines for Uterine<br>Fibroids | Туро |
|---|---|---|---|
| 26 | 7.8.1.1Primary Analysis | 7.8.1.1Primary Analysis | Туро |
| | If the lower bound of the 95%CI is greater or equal to the non-inferiority margin of 15%,, then non-inferiority of TAK-385 40mg to leuprorelin will be concluded. | If the lower bound of the 95%CI is greater or equal to the non-inferiority margin of -15%, then non-inferiority of TAK-385 40mg to leuprorelin will be concluded. | |
| 27 | 7.8.1.4Examination of Subgroups | 7.8.1.4Examination of Subgroups | Removed based on blind review |
| | Cervical Fibroid[Yes, No] | removed | |
| 28 | 7.8.2.1PBAC Score | 7.8.2.1PBAC Score | Specify the detail |
| | For each variable, frequency will be summarized by treatment group. The point estimate and 2-sided 95% confidence interval of the difference in the percentage will be calculated between TAK-385 40 mg group and leuprorelin group, using FM method. | For each variable, frequency will be summarized by treatment group. The point estimate and 2-sided 95% confidence interval of the difference in the percentage will be calculated between TAK-385 40 mg group and leuprorelin group, using FM method with the non-inferiority margin of -15%. The confidence interval will be presented in a descriptive manner and not for the purpose of statistical inference. | description how to calculate CI using FM method, based on the comment. |
| 29 | 7.8.2.3Hemoglobin | 7.8.2.3Hemoglobin HGB at Baseline (g/dL)[Min<= - <12, 12<= - <=Max] | Added based on blind review |
| 32 | | Section 7.8.3.4 was newly added. | Added based on the comment. |

| 42 | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | Modified based on blind review |
|---|---|---|---|
| | For each variable, summaries (1) and (2) will be provided by treatment group. | For each variable except T score, summaries (1), (3), and (4) will be provided by treatment group. | |
| 42 | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | Modified based on blind review |
| | For T score, summary (3) will be provided by treatment group. | For T score, summary (2), (3), (4), and (5) will be provided by treatment group. | |
| 42 | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | 7.11.5.1Bone Mineral<br>Density and Biochemical<br>Bone Metabolism Markers | Modified based on blind review |
| | Descriptive statistics for observed values for each visit and changes from baseline will be provided. | Descriptive statistics for observed values for each visit and percent changes from baseline will be provided. | |
| 42 | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | Modified based on blind review |
| | | (2)Summary of Parameters<br>and Change from Baseline<br>by Visit | |
| | | Descriptive statistics for observed values for each visit and changes from baseline will be provided. | |
| 43 | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | 7.11.5.1Bone Mineral Density and Biochemical Bone Metabolism Markers | Modified based on blind review |
| | | (4)Mean Plot with Standard<br>Deviations | |

| | | For T score, mean of observed values and changes from baseline will be plotted by visit. | |
|---|---|---|---|
| | | For other variables, mean of observed values and percent changes from baseline will be plotted by visit. | |
| 45 | Appendix 1. Criteria for Markedly Abnormal Values For each parameter, all evaluable data (i.e., nonmissing and acceptable according to the Handling Rules for Analysis Data) obtained up to Follow-up Day 14 will be classified as a MAV or not. | Appendix 1. Criteria for Markedly Abnormal Values For each parameter, all evaluable data (i.e., nonmissing and acceptable according to the Handling Rules for Analysis Data) obtained up to Follow-up Day 42 will be classified as a MAV or not. | Modified to be accordance with CCT-001 study. |
| 46 | Appendix 1. Criteria for<br>Markedly Abnormal Values<br>Pulse (bpm) | Appendix 1. Criteria for<br>Markedly Abnormal Values<br>Pulse Rate (bpm) | Туро |
| 46 | Appendix 1. Criteria for<br>Markedly Abnormal Values<br>Body Temperature (°C) | Appendix 1. Criteria for<br>Markedly Abnormal Values<br>Body temperature (°C) | Туро |
| 48 | Appendix 2. Criteria for Elevated Liver Enzyme All evaluable data (ie, nonmissing and acceptable according to the Handling Rules for Analysis Data) obtained up to Follow-up Day 14 will be used to determine whether each criteria for elevated liver enzyme in the table below is met or not. | Appendix 2. Criteria for Elevated Liver Enzyme All evaluable data (ie, nonmissing and acceptable according to the Handling Rules for Analysis Data) obtained up to Follow-up Day 42 will be used to determine whether each criteria for elevated liver enzyme in the table below is met or not. | Modified to be accordance with CCT-001 study. |
| 52 | Appendix 3. UFS-QoL<br>Scoring Manual | Appendix 3. UFS-QoL<br>Scoring Manual | Modified based on blind review |

| | Transformed Score =((Actual raw score – lowest possible raw score)/(Possible raw score range))*100 | Transformed Score =((Actual raw score – lowest possible raw score)/(Possible raw score range))*100 (rounded to the nearest integer) | |
|---|---|---|---|
| 53 | Appendix 3. UFS-QoL<br>Scoring Manual | Appendix 3. UFS-QoL<br>Scoring Manual | Modified based on blind review |
| | Transformed Score =((Highest possible score – Actual raw score)/(Possible raw score range))*100 | Transformed Score =((Highest possible score – Actual raw score)/(Possible raw score range))*100 (rounded to the nearest integer) | |
| 54 | Appendix 4. WPAI Scoring Manual | Appendix 4. WPAI Scoring Manual | Modified based on blind review |
| | Multiply scores by 100 to express in percentages. | Multiply scores by 100 to express in percentages (rounded to the nearest integer). | |

# **8.0 REFERENCES**

Farrington C P, Manning G: Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference or non-unity relative risk. Statistics in Medicine 1990; 9: 1447-1454.